CLINICAL TRIAL: NCT07384806
Title: The Effect of Functional Training on Speed, Balance, and Functional Capacity in Adolescent Table Tennis Players: A Randomized Controlled Trial
Brief Title: Functional Training in Adolescent Table Tennis
Acronym: FT in Adolesce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alirıza Han Civan (Other)
Responsible Party: Sponsor-Investigator, Alirıza Han Civan, Dr, Karabuk University
Organization: Karabuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-77192459-050.99-381871
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Functional Training in Adolescent Table Tennis Players
Keywords: Functional Training; Table Tennis; Adolescents; Physical Performance; Agility; Balance; Speed; Functional Movement Screen; Vertical Jump; Multi-Joint Exercises

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial evaluating the effects of functional training on physical performance in adolescent table tennis players. Participants are randomly allocated to one of three groups: Functional Training, Conventional Training, or Control. Measurements are taken at pre-test, mid-test, and post-test timepoints.
Masking Description: No masking was applied in this study. Participants, investigators, and outcome assessors were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional Training Group (Experimental): Eight-week functional training program focusing on flexibility, agility, speed, balance, and movement quality. Training is performed three times per week alongside regular table tennis practice.
  Interventions: Behavioral: Functional Training
- Conventional Training Group (Active Comparator): Participants perform conventional table tennis training for eight weeks following standard club routines.
  Interventions: Behavioral: Conventional Training
- Control Group (No Intervention): Participants continue their usual routine table tennis training without any additional intervention.

INTERVENTIONS:
Behavioral: Functional Training — Eight-week functional training program focusing on flexibility, agility, speed, balance, and movement quality. Training is performed three times per week alongside regular table tennis practice.
  Arms: Functional Training Group
Behavioral: Conventional Training — Standard table tennis training performed three times per week for eight weeks without additional functional exercises.
  Arms: Conventional Training Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of an eight-week functional training program on physical performance parameters in adolescent table tennis players. Functional training involves multi-joint and multi-plane exercises designed to improve movement quality, strength, balance, and coordination.

Thirty adolescent table tennis players will be randomly assigned to one of three groups: Functional Training, Conventional Training, or Control (routine training). The Functional Training group will perform a structured functional exercise program in addition to regular table tennis training, while the Conventional Training group will continue standard training routines. The Control group will maintain regular practice only.

Physical performance variables including flexibility, agility, speed, vertical jump performance, functional movement patterns, and balance will be assessed before, during, and after the intervention period.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to examine the effects of an eight-week functional training program on physical performance in adolescent table tennis players. Functional training focuses on multi-joint, multi-planar exercises aimed at improving movement efficiency, balance, strength, and neuromuscular coordination.

Thirty adolescent table tennis players aged 12-16 years with at least three years of training experience will be recruited and randomly allocated to one of three groups: Functional Training, Conventional Training, or Control. The Functional Training group will perform a structured exercise program consisting of dynamic, whole-body movements designed to enhance agility, balance, speed, and movement quality. Training sessions will be conducted three times per week for eight weeks in addition to regular table tennis practice.

The Conventional Training group will continue standard technical and tactical training without additional functional exercises. The Control group will maintain routine training only.

Outcome measures will be collected at baseline, mid-intervention, and post-intervention. Assessments will include flexibility, agility, sprint speed, vertical jump performance, Functional Movement Screen scores, and static and dynamic balance measures. Outcome measures will be collected at baseline, mid-intervention, and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescent table tennis players aged 12-18 years.
* Actively training and competing in table tennis for at least 2 years.
* Participating in at least 3 training sessions per week.
* Free from injury or medical conditions affecting physical performance.
* Voluntarily consent to participate in the study (parental consent required for minors).

Exclusion Criteria:

* Any musculoskeletal injury, neurological disorder, or medical condition affecting training or performance.
* Participation in another structured training program during the study period.
* Non-compliance with study protocol or inability to attend scheduled sessions.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-11-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-03 (Actual)

PRIMARY OUTCOMES:
Overall Physical Performance Score | Baseline (pre-test), mid-intervention (week 4), and post-intervention (week 8)
  Overall physical performance will be assessed using a battery of standardized physical performance tests including flexibility, agility, speed, vertical jump height, balance, and Functional Movement Screen (FMS).
  Flexibility: Sit-and-Reach Test (cm; higher values indicate better flexibility) Agility: T-test (seconds; lower values indicate better performance) Speed: 10-meter sprint test (seconds; lower values indicate better performance) Vertical Jump: Countermovement jump height (cm; higher values indicate better performance) Balance: Static and dynamic balance tests (test-specific scoring; higher scores indicate better balance) Functional Movement Screen (FMS): Composite score ranging from 0 to 21, with higher scores indicating better movement quality

SECONDARY OUTCOMES:
Flexibility (Sit-and-Reach Test) | Baseline (pre-test), mid-intervention (week 4), and post-intervention (week 8)
  Flexibility will be assessed using a sit-and-reach test that measures the flexibility of the hamstring and lower back muscles.
  Measurement: Sit-and-reach Test Unit: centimeters (cm) Range: Typically 0-50 cm Direction: Higher scores indicate better flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Alirıza Han Civan, Dr, Principal Investigator — Karabük Üniversitesi Hasan Doğan Spor Bilimleri Fakültesi Spor Yöneticiliği Bölümü
Locations (1):
- Karabük University, Karabük, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared in this study. Study data were analyzed solely by the research team and will not be shared with third parties to protect participant confidentiality.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT07384806/Prot_SAP_000.pdf